CLINICAL TRIAL: NCT03756584
Title: Probing TBS-induced Neural Plasticity and Associated Effects on Learning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Georg Kranz (Other)
Responsible Party: Sponsor-Investigator, Dr Georg Kranz, Principal Investigator, The Hong Kong Polytechnic University
Organization: The Hong Kong Polytechnic University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 1-ZVN9
Record Dates: First submitted 2018-11-22; First posted 2018-11-28 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Healthy
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: single-blind parallel-group crossover design
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent theta-burst stimulation (Experimental): iTBS will be performed on the left lateral parietal cortex
  Interventions: Device: Theta-burst stimulation
- Control stimulation (Active Comparator): iTBS will be performed on the vertex
  Interventions: Device: Theta-burst stimulation

INTERVENTIONS:
Device: Theta-burst stimulation — iTBS comprises 3-pulse 50-Hz bursts, applied every 200 ms (at 5 Hz) as described previously (Huang, Edwards et al. 2005) and consists of 2-second trains with an inter-train-interval of 8 seconds. We will repeat trains (30 pulses; 10 bursts) for 20 times to reach a total number of 600 pulses per session (3x10x20)
  Other Names: Transcranial Magnetic Stimulation

SUMMARY:
Recent animal research indicates that excitatory brain stimulation opens a time window of increased neural plasticity that permits remodeling of neural representations. Repetitive transcranial magnetic stimulation (rTMS) may thus facilitate learning of new associations by reducing proactive interference but human research is missing. Therefore, it is the aim of this study to investigate the effects of intermittent theta-burst stimulation (iTBS), a potent form of excitatory brain stimulation, on associative memory. Twenty right handed healthy participants will receive 3 minutes of iTBS or sham stimulation of the left lateral parietal cortex after memorizing a set of 20 face-word associations. Recall capacity will be tested directly before and after stimulation. Participants will then learn a new combination of associations using the same set of stimuli, followed by an evaluation of their recall capacity. It is hypothesized that iTBS compared to sham stimulation will reduce recall capacity directly after the stimulation but increase recall capacity of the newly learned associations due to reduced proactive interference. This study may not only pave the way towards a new understanding of the mechanism of action of brain stimulation, but can also help in developing new treatment strategies for neuropsychiatric disorders.

ELIGIBILITY:
Inclusion Criteria:

* education level of primary six or above
* right-handedness
* normal or corrected-to-normal vision

Exclusion Criteria:

* seizures in medical history
* current or past psychiatric disorders or severe internal or neurological illness
* common TMS exclusion criteria
* substance abuse or dependence
* intake of medication that is known to affect the excitation threshold

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2019-03-03 (Actual); Primary Completion 2020-12-03 (Actual); Study Completion 2020-12-03 (Actual)

PRIMARY OUTCOMES:
Change in recall capacity | Change from baseline to directly after stimulation (~6 min after baseline)
  Change in the number of correct associations of a face-word association memory test

CONTACTS AND LOCATIONS:
Overall Officials: Georg S Kranz, PhD, Principal Investigator — Department of Rehabilitation Sciences
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Behavioral data may be shared with other researchers